CLINICAL TRIAL: NCT00747955
Title: Evaluation of Assessments of Motor Performance, Physical Impairments and Functional Abilities
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 080205; 08-CC-0205
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-04-07

CONDITIONS: Healthy Volunteers
Keywords: Human Performance; Physical Disability; Functional Outcome Measures; Health Volunteer; HV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will evaluate new assessment tools and equipment and new ways of using existing tools and equipment in the NIH Clinical Center s Rehabilitation Medicine Department in order to maximize patients function. The Department assesses and treats NIH patients with chronic pain, problems in walking or getting around, activities of daily living, performing tasks needed for jobs or hobbies, communicating and chewing and swallowing.

Children and adults of all ages with disabilities and healthy normal volunteers may be eligible for this study.

The following kinds of assessments are evaluated in this study:

Assessments of Impairments

Impairments are problems such as loss of movement, weakness or loss of sensation. Assessments may include measurements of range of motion, strength, sensation, pain, joint stability or mobility, joint angles, limb and girth, gait, exercise tolerance, stamina, or ultrasound imaging of muscle and swallowing function.

Assessments of Function and Performance

Functional and performance assessments look at how well subjects perform actions, such as walking or getting around, dressing, or preparing meals. They may include evaluations of activities of daily living, leisure activities, fatigue, vocational activity, school activity, coping skills, and quality of life. The assessments may be done by questionnaires or interviews and by watching subjects perform the activities.

Assessments of Treatment Techniques

Treatment techniques are assessed by evaluating methods and equipment used to treat patients with impairments or problems with function. They may evaluate, for example, the use of heat, cold, strengthening exercises, fitness exercises, TENS units, splinting and orthotics, or shoe modifications.

DETAILED DESCRIPTION:
Objective

The objective of the protocol is to provide framework in which clinicians in the Department of Rehabilitation Medicine (RMD) can serve the clinical needs of patients and the intramural clinical research needs of NIH investigators by maintaining state of the art expertise in the functional assessment of persons with disabilities and investigating new equipment, methodologies and/or techniques for functional assessment.

Study Population

We intend to study a total of 500 healthy volunteers and 500 subjects with disabilities, including those enrolled in NIH intramural research protocols.

Design

The study will consist of individual projects designed designed by RMD staff including one or more of the associate investigators. The individual projects will be relatively small and designed to test the reliability, reproducibility, efficiency, feasibility, sensitivity, specificity, tolerability, validity and/or precision of physical medicine and rehabilitation assessment equipment, devices and clinical evaluations of impairment, disability, and/or function.

Outcome Measures

The specific outcome measure(s) will be chosen to meet the goals of the individual project and will generally include one or more of the following:

i. Subjective assessment by the participant of the test, device, or evaluation based on written evaluation tools.

ii. Comparisons to established evaluations or equipment designed to assess similar areas of function, including concurrent validity analyses.

iii. Subjective assessment by clinicians using the test, device or evaluation, based on written evaluation tools.

iv. Feasibility assessments, including the time required for participants to perform tests, time for clinicians to evaluate the results of the tests, and/or prepare reports of the results of tests.

v. Assessments of reliability and/or stability of the technique used, including statistical tests of coefficients of variability.

vi. Assessments of tolerance of tests, including measures such as vital signs or elements of a physical examination.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion criteria for subjects with disabilities

To participate in projects in this study, subjects with disabilities must:

* have a disability appropriate to the measure being assessed
* be clinically stable and medically able to tolerate the measure to be evaluated in a specific project in which they are to be enrolled
* be an adult able to give informed consent or, if a minor, have a parent/guardian able to provide informed consent
* be at least 2 years of age, with no upper age limit

Inclusion criteria for healthy volunteers

To participate in projects in this study, healthy volunteers must:

* be an adult able to provide informed consent or, if a minor, have a parent/guardian able to provide informed consent
* be in good general health and have no disability
* be able medically able to tolerate the measure to be evaluated in the specific project in which they are to be enrolled
* be at least 2 years of age, with no upper age limit

EXCLUSION CRITERIA:

Exclusion criteria for subjects with disabilities

* Have limitations relating to their disability that could result in pain or injury on attempt to use the device or participate in the measure being evaluated in the specific project in the study
* Are unable to understand the instructions required to safely use the device or participate in the measure being evaluated
* Have a medical or other device in or on their body which may interfere the research assessments.
* Have a medical or other device in or on their body that places them at increased risk from use of any device to be evaluated, based on manufacturer s recommendations or accepted medical literature
* Have any medical condition which contraindicates use of the specific device to be evaluated, based on manufacturer s recommendations or accepted medical literature.

Exclusion criteria for healthy volunteers

* Are discovered to have a previously undiagnosed impairment or disability in the domain to be evaluated by the device or measure to be used in the specific project in the study
* Are unable to understand the instructions required to safely use the device or participate in the measure being evaluated.
* Have a medical or other device in or on their body which may interfere the research assessments.
* Have a medical or other device in or on their body that places them at increased risk from use of any device to be evaluated, based on manufacturer s recommendations or accepted medical literature
* Have any medical condition which contraindicates use of the specific device to be evaluated, based on manufacturer s recommendations or accepted medical literature
* RMD special volunteers, employees and contractors will not be able to participate in this protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-08-28; Study Completion 2017-04-07

PRIMARY OUTCOMES:
To evaluate use of clinical assessments/equipment | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Paul, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States